CLINICAL TRIAL: NCT00808301
Title: Multicentre Clinical Trial on Oat Products in the Treatment of Coeliac Disease in Children
Brief Title: Oat Products in the Treatment of Coeliac Disease in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heinz Italia SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLA-07-01
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Clinical and Nutritional Safety.
Keywords: Coeliac disease; Oat
MeSH Terms: conditions — Celiac Disease; Gyrate Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A/B (Other): This is a cross-over design, i.e. each patient is treated with either oat or control products in different times.
  Interventions: Other: Gluten-free products

INTERVENTIONS:
Other: Gluten-free products — Gluten-free bakery products containing oatmeal.
  Other Names: BiAglut

SUMMARY:
In many Northern European countries oat-based products have been used in the dieto-therapy of coeliac disease for many years.

The purpose of this study is to evaluate clinical tolerance and liking of gluten-free products containing oatmeal from a specific oat variety (not contaminated with gluten) in a sample of Italian celiac patients in pediatric age.

DETAILED DESCRIPTION:
Several clinical trials have demonstrated that most celiac patients, both of pediatric and of adult age, can take medium-high quantity of oat (50-100 g/day), without any negative clinical effects.

In a small number of cases intestinal dyspeptic disorders, especially meteorism, can be observed, particularly during the first weeks of oat intake. They are generally without clinical significance because they are a consequence of the increased fibre intake.

There are only few cases of "true" oats intolerance. The addition of oat improves the nutritional quality of the gluten-free diet, particularly due to the increased intake of fibre and some oligoelements (iron, zinc, tiamin, pholates) and expands the spectrum of food choices.

In many Northern European countries oat-based products have been used in the dieto-therapy of coeliac disease for many years.

For the oat-based product to be considered suitable in the dieto-therapy of coeliac disease, the absence of gluten contamination and possibly the origin from a variety of oat which is without traces of gluten cross-reactive peptides must be guaranteed.

The purpose of this study is to evaluate clinical tolerance and liking of gluten-free products containing oatmeal from a specific oat variety (not contaminated with gluten) in a sample of Italian celiac patients in pediatric age.

ELIGIBILITY:
Inclusion Criteria: the study will include patients aged between 4 and 14, under treatment with a gluten-free diet for coeliac disease (bioptic diagnosis) for at least two years.

Exclusion Criteria:

diagnosis not confirmed by intestinal biopsy, cases with little adherence to the treatment (anti-tTG positive at basal evaluation), cases of potential coeliac disease (completely normal mucous membrane), cases with an associated sieric IgA deficit, cases with associated diseases (es. diabetes type 1).

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-07 (Actual); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Clinical safety through serological markers of coeliac disease and intestinal wall integrity, clinical and bioumoral parameters of nutrition status, frequency and clinical type of dyspeptic disorders or other adverse reactions. | Controls at recruiting, after 3, 6, 9, 12, 15 months from the beginning of the study.

SECONDARY OUTCOMES:
Liking of gluten-free products containing oatmeal is evaluated through a product liking questionnaire. | Product liking questionnaire after 6 months and 15 months from the beginning of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Catassi, Prof., Principal Investigator — Università Politecnica delle Marche - Clinica Pediatrica - Ancona; Ruggiero Francavilla, Dr., Principal Investigator — Ospedale Policlinico Consorziale, Clinica Pediatrica "B.Trambusti" - Bari; Klaus Pittschieler, Prof., Principal Investigator — Ospedale Centrale di Bolzano; Basilio Malamisura, Prof., Principal Investigator — Ospedale Civile "S. Maria Incoronata dell'Olmo" - Cava de' Tirreni (SA); Roberto Panceri, Dr., Principal Investigator — Azienda Ospedaliera "San Gerardo" - Monza; Maria Barbato, Prof., Principal Investigator — Azienda Policlinico Umberto I, Roma; Mario La Rosa, Prof., Principal Investigator — Azienda Ospedaliero-Universitaria Policlinico Vittorio Emanuele, Catania
Locations (7):
- Italy (7):
  - Azienda Ospedaliero-Universitaria "Policlinico Vittorio Emanuele", Catania, CT
  - Ospedale Civile "S. Maria Incoronata dell'Olmo", Divisione di Pediatria, Cava de' Tirreni, Salerno
  - Università Politecnica delle Marche, Clinica Pediatrica, Ancona
  - Ospedale Policlinico Consorziale, Clinica Pediatrica "B.Trambusti", Bari
  - Ospedale Centrale, Divisione di Pediatria, Bolzano
  - Azienda Ospedaliera "San Gerardo", Clinica Pediatrica, Monza
  - Azienda Policlinico "Umberto I" - Dip. di Pediatria - UOC di Gastroenterologia ed Epatologia Pediatrica, Roma

REFERENCES:
- [Background] Catassi C. The world map of celiac disease. Acta Gastroenterol Latinoam. 2005;35(1):37-55. No abstract available. English, Spanish. PMID 15954735
- [Background] Fasano A, Catassi C. Current approaches to diagnosis and treatment of celiac disease: an evolving spectrum. Gastroenterology. 2001 Feb;120(3):636-51. doi: 10.1053/gast.2001.22123. PMID 11179241
- [Background] Reunala T, Collin P, Holm K, Pikkarainen P, Miettinen A, Vuolteenaho N, Maki M. Tolerance to oats in dermatitis herpetiformis. Gut. 1998 Oct;43(4):490-3. doi: 10.1136/gut.43.4.490. PMID 9824575
- [Background] Hoffenberg EJ, Haas J, Drescher A, Barnhurst R, Osberg I, Bao F, Eisenbarth G. A trial of oats in children with newly diagnosed celiac disease. J Pediatr. 2000 Sep;137(3):361-6. doi: 10.1067/mpd.2000.109003. PMID 10969261
- [Background] Janatuinen EK, Kemppainen TA, Julkunen RJ, Kosma VM, Maki M, Heikkinen M, Uusitupa MI. No harm from five year ingestion of oats in coeliac disease. Gut. 2002 Mar;50(3):332-5. doi: 10.1136/gut.50.3.332. PMID 11839710
- [Background] Storsrud S, Olsson M, Arvidsson Lenner R, Nilsson LA, Nilsson O, Kilander A. Adult coeliac patients do tolerate large amounts of oats. Eur J Clin Nutr. 2003 Jan;57(1):163-9. doi: 10.1038/sj.ejcn.1601525. PMID 12548312
- [Background] Lundin KE, Nilsen EM, Scott HG, Loberg EM, Gjoen A, Bratlie J, Skar V, Mendez E, Lovik A, Kett K. Oats induced villous atrophy in coeliac disease. Gut. 2003 Nov;52(11):1649-52. doi: 10.1136/gut.52.11.1649. PMID 14570737
- [Background] Hogberg L, Laurin P, Falth-Magnusson K, Grant C, Grodzinsky E, Jansson G, Ascher H, Browaldh L, Hammersjo JA, Lindberg E, Myrdal U, Stenhammar L. Oats to children with newly diagnosed coeliac disease: a randomised double blind study. Gut. 2004 May;53(5):649-54. doi: 10.1136/gut.2003.026948. PMID 15082581
- [Background] Arentz-Hansen H, Fleckenstein B, Molberg O, Scott H, Koning F, Jung G, Roepstorff P, Lundin KE, Sollid LM. The molecular basis for oat intolerance in patients with celiac disease. PLoS Med. 2004 Oct;1(1):e1. doi: 10.1371/journal.pmed.0010001. Epub 2004 Oct 19. PMID 15526039
- [Background] Holm K, Maki M, Vuolteenaho N, Mustalahti K, Ashorn M, Ruuska T, Kaukinen K. Oats in the treatment of childhood coeliac disease: a 2-year controlled trial and a long-term clinical follow-up study. Aliment Pharmacol Ther. 2006 May 15;23(10):1463-72. doi: 10.1111/j.1365-2036.2006.02908.x. PMID 16669961
- [Background] Peraaho M, Collin P, Kaukinen K, Kekkonen L, Miettinen S, Maki M. Oats can diversify a gluten-free diet in celiac disease and dermatitis herpetiformis. J Am Diet Assoc. 2004 Jul;104(7):1148-50. doi: 10.1016/j.jada.2004.04.025. PMID 15215774
- [Background] Garsed K, Scott BB. Can oats be taken in a gluten-free diet? A systematic review. Scand J Gastroenterol. 2007 Feb;42(2):171-8. doi: 10.1080/00365520600863944. PMID 17327936
- [Background] Storsrud S, Hulthen LR, Lenner RA. Beneficial effects of oats in the gluten-free diet of adults with special reference to nutrient status, symptoms and subjective experiences. Br J Nutr. 2003 Jul;90(1):101-7. doi: 10.1079/bjn2003872. PMID 12844381
- [Background] Thompson T. Gluten contamination of commercial oat products in the United States. N Engl J Med. 2004 Nov 4;351(19):2021-2. doi: 10.1056/NEJM200411043511924. No abstract available. PMID 15525734
- [Background] Hernando A, Mujico JR, Juanas D, Mendez E. Confirmation of the cereal type in oat products highly contaminated with gluten. J Am Diet Assoc. 2006 May;106(5):665; discussion 665-6. doi: 10.1016/j.jada.2006.03.024. No abstract available. PMID 16647318
- [Background] Hollen E, Hogberg L, Stenhammar L, Falth-Magnusson K, Magnusson KE. Antibodies to oat prolamines (avenins) in children with coeliac disease. Scand J Gastroenterol. 2003 Jul;38(7):742-6. doi: 10.1080/00365520310003156. PMID 12889560
- [Background] Fasano A, Not T, Wang W, Uzzau S, Berti I, Tommasini A, Goldblum SE. Zonulin, a newly discovered modulator of intestinal permeability, and its expression in coeliac disease. Lancet. 2000 Apr 29;355(9214):1518-9. doi: 10.1016/S0140-6736(00)02169-3. PMID 10801176
- [Derived] Lionetti E, Gatti S, Galeazzi T, Caporelli N, Francavilla R, Cucchiara S, Roggero P, Malamisura B, Iacono G, Tomarchio S, Kleon W, Restani P, Brusca I, Budelli A, Gesuita R, Carle F, Catassi C. Safety of Oats in Children with Celiac Disease: A Double-Blind, Randomized, Placebo-Controlled Trial. J Pediatr. 2018 Mar;194:116-122.e2. doi: 10.1016/j.jpeds.2017.10.062. PMID 29478494